CLINICAL TRIAL: NCT06865040
Title: Perioperative Inhaled Therapy in Carcinological Thoracic Surgery in Patients at High Risk of Postoperative Pulmonary Complications
Acronym: TICTAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2023_843_0151
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Surgery; Postoperative Pulmonary Complications (PPCs)
Keywords: Thoracic surgery; postoperative pulmonary complications; Inhaled therapy; bronchodilators; B2 mimetics
MeSH Terms: interventions — Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Administration in the interventional arm of long-acting inhaled ß-2 mimetics:
  FORMOTEROL FUMARATE 12 µg pwd inhalation capsule (FORMOTEROL VIATRIS®), taken twice a day intraoperatively from Day-2 to Day 7.
  Interventions: Drug: Formoterol Fumarate 12 mcg (Foradil Aerolizer)
- control group (Sham Comparator): The trial was conducted as an open-label study for the control group.
  Interventions: Other: Usual treatment

INTERVENTIONS:
Drug: Formoterol Fumarate 12 mcg (Foradil Aerolizer) — Administration in the interventional arm of long-acting inhaled ß-2 mimetics:
  FORMOTEROL FUMARATE 12 µg pwd inhalation capsule (FORMOTEROL VIATRIS®), taken twice a day intraoperatively from Day-2 to Day 7.
  Arms: experimental group
Other: Usual treatment — usual treatment
  Arms: control group

SUMMARY:
The objective of the study is to evaluate, in a clinical trial, the efficacy of peri operative administration of long-acting inhaled ß-2 mimetics on the occurrence of postoperative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* Lung cancer eligible for surgical management by lung resection (non-small cell lung carcinoma = NSCLC) by any route
* Naïve to long-term inhaled bronchodilator therapy
* High risk of post-operative pulmonary complications (Pre-operative FEV1 < 80%)

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Emergency surgery
* Patient with a physiological status of WHO IV or ASA ≥ IV
* Asthma
* Patients treated with long-acting bronchodilators
* Severe heart failure (NYHA IV), unstable ischaemic heart disease (angina or recent infarction < 3 months), obstructive hypertrophic cardiomyopathy, subvalvular aortic stenosis, severe uncontrolled hypertension Recent stroke < 3 months
* High-grade unresponsive conductive disorders or unstable arrhythmia
* Thyrotoxicosis, pheochromocytoma
* Unbalanced diabetes
* Hypersensitivity to ß-2 mimetics or lactose
* Current participation in a trial of another drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of postoperative pulmonary complication | day 7
  Number of postoperative pulmonary complications (PPC) at day 7 after a thoracic surgery for lung resection

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No